CLINICAL TRIAL: NCT00000765
Title: Pilot Study to Evaluate the Efficacy of Zidovudine in Preventing CD4+ Lymphocyte Decline in Patients With Primary HIV Infection. (One Treatment Arm Receives Placebo)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: DATRI 002; 11733 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety and efficacy of early treatment with zidovudine for preventing a decline in CD4+ lymphocyte counts in patients with primary HIV infection. To determine the natural history of virologic and immunologic changes in primary HIV infection.

Previous studies indicate that intervention with zidovudine during primary HIV infection could reduce the initial viral burden and subsequent decline in immune functions, and could prolong not only the time to development of AIDS but also the time to initiation of chronic antiretroviral therapy.

DETAILED DESCRIPTION:
Previous studies indicate that intervention with zidovudine during primary HIV infection could reduce the initial viral burden and subsequent decline in immune functions, and could prolong not only the time to development of AIDS but also the time to initiation of chronic antiretroviral therapy.

Patients are randomized to receive either zidovudine or placebo daily for 24 weeks. Patients are followed until development of an AIDS-related opportunistic infection or malignancy. After week 24, patients meeting standard prescribing criteria may start FDA-approved anti-HIV therapies. After study week 48, patients may co-enroll on another clinical trial to receive experimental therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Medications for nausea, vomiting, analgesia, or anxiety.

Patients must have:

* Asymptomatic or symptomatic primary HIV infection, plus one of the following two criteria:

  1. p24 antigenemia documented within 1 month prior to study entry and either HIV enzyme immunoassay (IA) negative or HIV IA positive with Western blot negative/indeterminate, within 1 month prior to study entry.
  2. Documented seroconversion within 1 month prior to study entry and Western blot negative/indeterminate.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following condition are excluded:

* poor venous access.

Concurrent Medication:

Excluded:

* Chronic steroid use.
* Immunomodulators.
* Myelosuppressive agents.
* Other antiretroviral agents or experimental therapies (NOTE: FDA-approved therapies permitted in patients who qualify after week 24; experimental therapies permitted after study week 48).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Niu, Study Chair; H Standiford, Study Chair
Locations (9):
- United States (9):
  - Cedars Sinai Med Ctr, Los Angeles, California
  - Palo Alto Veterans Administration Med Ctr, Palo Alto, California
  - Broward Gen Med Ctr, Fort Lauderdale, Florida
  - Univ of Illinois, Chicago, Illinois
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas

REFERENCES:
- [Background] Holodniy M, Niu M, Bethel J, Standiford H, Schnittman S. A pilot study to evaluate the efficacy of zidovudine (ZDV) versus placebo in primary HIV infection (DATRI 002): a preliminary analysis. Int Conf AIDS. 1996 Jul 7-12;11(Program Supplement):26 (abstract no LBB6022)